CLINICAL TRIAL: NCT06643624
Title: Effects of Vision Training on Sportive Performance in Professional Wrestlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tuğba Kuru Çolak, Principal İnvestigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MU-SBE-FTR-MŞE-01
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Health Individuals
Keywords: vision training; wrestling; sportive performance

STUDY DESIGN:
Intervention Model Description: There are two groups: one group is the control group and the other is the vision training group, in which vision training is applied.
Who Masked: Participant
Masking Description: the athletes participating in the study did not know which group they were in, whether the other group received the same training, or if they did, what kind of procedure was applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The athletes in the control group continued their routine training program. no vision training program was applied to the athletes in this group.
  Interventions: Other: Routine Training Program
- Vision Training Group (Experimental): In addition to their routine training program, the athletes in the vision training group were subjected to a vision training program administered by a physiotherapist, which gradually increased in duration over 8 weeks.
  Interventions: Other: Vision Training Program; Other: Routine Training Program

INTERVENTIONS:
Other: Vision Training Program — Vision training (experimental) group; vision training program was applied in addition to routine training programs. For 8 weeks, 5 sessions per week for a total of 40 sessions of vision training were applied by a physiotherapist. In the first 2 weeks, each movement was applied for 1 minute for a total of 10 minutes. In the 3rd week, each movement was practiced for 1.5 minutes for a total of 15 minutes. In weeks 4-8, each movement was performed for 2 minutes each for a total of 20 minutes.
  Arms: Vision Training Group
Other: Routine Training Program — All athletes performed their routine training for wrestling 6 days a week.

SUMMARY:
This study examines the effects of vision training on the sportive performance of professional wrestlers. In wrestling, rapid decision making, timely opponent detection and effective execution of strategic moves are highly dependent on visual perception skills. In this context, our study investigated how vision training improves wrestlers' sportive performance and neck proprioception.

DETAILED DESCRIPTION:
This study examines the effects of vision training on the sportive performance of professional wrestlers. In wrestling, rapid decision making, timely opponent detection and effective execution of strategic moves are highly dependent on visual perception skills. In this context, our study investigated how vision training improves wrestlers' sportive performance and neck proprioception.

Before the study, ethical approval was obtained from Marmara University Faculty of Medicine Ethics Committee with the number 09.2022.1084. The study was started with 28 athletes from the Turkish Greco-Roman A National Team and was carried out on 27 athletes after one athlete in the control group was injured. The athletes who were examined by an ophthalmologist before the study, who did not have any visual problems and who did not have a history of surgical operation and / or injury that would adversely affect the balance in the last 6 months were randomly divided into 2 groups. The 14-member vision training group was subjected to a vision training program that included eye exercises accompanied by a physiotherapist for 5 sessions per week in addition to their routine training for 8 weeks, while the control group continued their routine training. Performance measurements were performed in both groups at the beginning of the study, in the middle of the training (week 4.), at the end of the training (week 8.) and 4 weeks after the training (week12.). Performance evaluations; Wrestling Specific Shuttle Run, Squat-Bench Press Maximum Strength, The Mc-Gill Endurance (Flexion, Extension and Lateral Plank Endurance Tests), Pro-agility Agility, Stork Static Balance, Star Dynamic Balance (Anterior, Posterolateral and Posteromedial directions) and Neck Proprioception tests (cervical region flexion, extension, right lateral flexion, left lateral flexion, right rotation and left rotation). The measurement results were statistically evaluated both within and between groups. The effect of the training program on the visual training and control groups was compared in a time-dependent manner. The effect x time interaction was evaluated by ANOVA analysis.

ELIGIBILITY:
Inclusion Criteria:

* wrestling federation of turkey to take part in the national wrestling team Being between 18-35 years old

Exclusion Criteria:

* having any eye disease having any systemic disease balance problems has had an operation that affects vision and balance (e.g. anterior cruciate ligament) within the last 6 months history of any traumatic brain injury in the last 6 months any serious upper/lower extremity injury in the last three months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study was designed for the Greco-Roman wrestlers. And this style is only for men.
Enrollment: 27 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Neck (Cervical) Proprioception Assessment | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  With the help of a laser fixed on the head, neck flexion, extension, right & left lateral flexion, right & left rotation movements were performed. In the table opposite, the point at which the same movement occurred in each of the three repetitions was marked and measured. Measurements were averaged. After being formulated, it was evaluated whether the training improved the angular velocity and the person's neck movement position sense.

SECONDARY OUTCOMES:
Strength (Anaerobic) Test (number of rounds): Wrestling Specific Shuttle Test | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  This test, which was developed methodologically to evaluate the anaerobic capacities of wrestling athletes with wrestling-specific movements, is an easily applicable test in the training facility (on the mat) and without the need for foreign or special equipment.. The test is based on wrestling-specific 4-directional movements (forward running, backward running, left lateral and right lateral running and is performed on a wrestling mat. Each movement is performed from the center of the mat to points four meters long and participants try to achieve as many repetitions as possible by continuously repeating the shuttle runs within a 3-minute period.
Maximal Strength Test (kg): Squat Test -Bench Press Test | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  1 repetition maximum (lRM) was assessed by squatting and bench press (lifting with arms upwards) to measure the maximum dynamic strength of the athletes. The highest load that the individual could lift to full extension of the knees was considered valid for the squat test and the highest load that the individual could lift to full extension of the elbows was considered valid for the BP test. The athletes were subjected to 3 trials with 3-5 minute intervals for each test.
Core Endurance Test (sec): The Mc-Gill Test | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  In this test, the duration of maintaining a certain position of the trunk flexion, extension and lateral plank muscles was examined.
Agility Test: Pro-Agility Test | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  In order for an athlete to initiate a forward movement, the body's center of mass must shift forward or the base of support must shift behind the center of mass by placing one foot back. Similarly, when asked to move laterally, the same principles apply (Frost et al., 2008). Either when initiating a lateral movement, the center of pressure needs to be shifted by bringing one foot closer to the other to be placed behind the body's center of mass relative to the intended direction of acceleration, or the body's center of mass needs to be shifted to the left or right. The pro-agility test, also known as 5-10-5, is widely used by many organizations and coaches as one of the gold standards for measuring athletes' ability to change direction, which is used to define agility.
Static Balance Test: Stork Test | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  The static balance of the individuals was evaluated with the one-leg stand test. With eyes open and arms by the hips, the individual was asked to stand on his/her dominant (preferred) foot for as long as he/she could without any help from anywhere. The mean values of the measurements made three times were taken and this time was recorded in seconds.
Dynamic Balance Test: Y Balance Test | *Measure-1: Week 0 *Measure-2: week 4 *Measure-3rd: week 8 *Measure-4th: week 12
  The dynamic balance assessment of the individuals was measured using the Y balance test. For the test setup, three tape measures were attached to the ground at an angle of 120 degrees. The individual was asked to stand on his preferred foot at the intersection point of these three tape measures and reach with his/her fingertip in three directions: anterior, posteromedial and posterolateral. During the test, care was taken to ensure that the individual's hands were on his/her waist and the heel of the foot on which the individual was standing did not lift off the ground. The test was repeated in cases where the individual lost balance or received support from the outstretched foot. In the Y balance test measurement, the test was repeated three times for each direction and the average was taken and recorded in centimeters. The value was then calculated by formulating the formula.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba KURU COLAK, Prof.Dr., Study Director — Marmara University
Locations (1):
- Turkısh Wrestling Federation Mersinli Ahmet Facilities, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No